CLINICAL TRIAL: NCT05168124
Title: Study to Determine the Effectiveness of Therapy Methods (acceptance Commitment Therapy, Micro Breaks) in Patients with Chronic Fatigue Syndrome/ Myalgic Encephalomyelitis
Brief Title: Effectiveness of Acceptance Commitment Therapy or Micro Breaks in Patients with Chronic Fatigue Syndrome/ Myalgic Encephalomyelitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Schiebler (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Sarah Schiebler, Senior Physician, Department of Consultation-Liaison-Psychiatry and Psychosomatic Medicine, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-00671
Record Dates: First submitted 2021-11-20; First posted 2021-12-23 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Fatigue Syndrome, Chronic
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acceptance Commitment Therapy for chronic fatigue (Active Comparator): ACT for chronic fatigue involves psychoeducation on the clinical picture of CFS/ME and teaching coping strategies for dealing with symptoms, most notably fatigue, postexertional malaise, unrestful sleep, cognitive decline, and orthostatic dysregulation. For this purpose, the therapy manual designed for generalized anxiety disorders is adapted to the needs of patients with CFS, i.e., the exercises and worksheets that teach the acceptance- and mindfulness-based techniques are adapted to the symptoms (fatigue, powerlessness, unrestful sleep, among others). In addition, value goals and scopes of action are defined, in which the individual stress limits of each participant are identified and taken into account. In addition, it is recommended that the participants move within their respective energy limits under the regular evaluation of activity and rest phases using a diary, as well as regularly apply study-specific interventions between the appointments of group therapy.
  Interventions: Behavioral: Acceptance Commitment Therapy for chronic fatigue
- Micro breaks in everyday life for chronic fatigue (Active Comparator): Micro breaks in everyday life (MBEL) includes restructuring the patients' daily routine in terms of how they organize their breaks. A therapy manual is developed for this purpose, which is divided into three phases. In the first phase, patients learn to allow or integrate regular MB of one to five minutes in their daily routine. Appropriate examples are used to show when and where MB can be incorporated and this is practiced at home over the first few weeks until a routine has been established. Patients are encouraged to keep a break diary. In the second phase, the MBs are filled in with content. MB can be designed differently, e.g., with physical activity of moderate or high intensity, with short breathing or relaxation exercises, with nutrition or even with doing nothing. In the third phase, an individual optimization of the design of breaks in everyday life follows and an expansion towards meaningful mental time-out, a combination of relaxation break and mental activation.
  Interventions: Behavioral: Micro breaks in everyday life for chronic fatigue
- Waiting Group (No Intervention)

INTERVENTIONS:
Behavioral: Acceptance Commitment Therapy for chronic fatigue — ACT was originally developed for the treatment of depression and anxiety. Recently, a single study investigated ACT as a therapeutic approach in CFS/ME and showed no negative effects on disease progression. ACT is characterized by acceptance- and mindfulness-based techniques, serves to promote acceptance and the development of new value goals, and can thereby open up new perspectives on life, which would be promising in terms of a reduction of symptom focus that seems to be a crucial effective factor for an improvement in exhaustion states. The intervention involves psychoeducation and teaching coping strategies for dealing with symptoms, most notably fatigue, postexertional malaise, unrestful sleep, cognitive decline, and orthostatic dysregulation. For this purpose, the therapy manual designed for anxiety disorders is adapted to the needs of patients with CFS, the exercises and worksheets that teach the acceptance- and mindfulness-based techniques are adapted to the symptoms.
  Arms: Acceptance Commitment Therapy for chronic fatigue
Behavioral: Micro breaks in everyday life for chronic fatigue — In terms of break design in the work context, research in recent years has increasingly focused on so-called "micro breaks" (MB) - mini breaks of one to five minutes in length. Transferred to mini breaks in everyday life (MBEL), there have been found fundamentally positive effects in terms of performance, vitality and well-being, which could also have a positive impact on the clinical picture of CFS/ME. However, practically no research results are yet available with regard to the implementation of MB in everyday life of patients with CFS/ME. The effects of MB, on the other hand, have been tested several times in everyday work settings and showed desirable effects on mood, attention, fatigue, vitality, performance, and well-being.
  Arms: Micro breaks in everyday life for chronic fatigue

SUMMARY:
Chronic fatigue syndrome/myalgic encephalomyelitis (CFS/ME) is a distinct disease entity with an estimated prevalence of 0.3-0.7% and more common in women (3:1 ratio). It can be diagnosed according to the Institute of Medicine (IOM) 2015 consensus definition using 3 major criteria and one of 2 minor criteria.

Diagnosis requires that the patient have the following three symptoms:

1. A substantial reduction or impairment in the ability to engage in pre-illness levels of occupational, educational, social, or personal activities that persists for more than 6 months and is accompanied by fatigue, which is often profound, is of new or definite onset (not lifelong), is not the result of ongoing excessive exertion, and is not substantially alleviated by rest,
2. Post-exertional malaise,* and
3. Unrefreshing sleep*

At least one of the two following manifestations is also required:

1. Cognitive impairment* or
2. Orthostatic intolerance

Note* Frequency and severity of symptoms should be assessed. The diagnosis of ME/CFS should be questioned if patients do not have these symptoms at least half of the time with moderate, substantial, or severe intensity.

Currently, individually tailored therapy with emphasis on cognitive behavioral therapy and graduated activity therapy is considered the therapy of first choice, although their effectiveness has been critically questioned in recent years. There are often frustrating treatment courses, a larger proportion of partial remissions, a significantly smaller proportion of full remissions and return to work.

The study aims to evaluate patients of the outpatient service for chronic fatigue at the Department of Consultation-Liaison Psychiatry and Psychosomatic Medicine, University Hospital Zurich, Switzerland, in the context of a group therapy for the treatment of CFS/ME in respect to the response to different, non-drug based therapeutic procedures and to gain knowledge about the effects of the therapy.

The study is a clinical comparative study of therapeutic procedures/interventions without the use of drugs or a medical product. The interventions are Acceptance Commitment Therapy (ACT) and Micro Breaks in Everyday Life (MBEL) adapted to CFS/ME. The collection of biological samples (saliva, blood) and health-related personal data (actigraphy, psychometric data from questionnaires) is associated with minimal risks and burdens.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis for CFS/ME
* Psychiatric clinical stability in the past 3 months:
* No diagnostic change to other categories of the International Classification of Diseases (ICD-10)
* No psychiatric inpatient treatments
* No psychiatric emergency treatments
* No suicide attempts
* Possession of internet access
* Sufficient skills to use electronic devices
* The willingness to engage in the described therapeutic procedures or interventions (ACT, MBEL)

Exclusion Criteria:

* Insufficient knowledge of German
* Severe psychiatric disorders (e.g. personality and posttraumatic stress disorders, dissociative and psychotic disorders, intelligence reduction, untreated attention deficit hyperactivity disorder) and acute suicidal tendencies
* Untreated or severe internal medicine disorders e.g., thyroid dysfunction, central and obstructive sleep apnea syndrome (i.e., apnea-hypopnea index >15 and/or "high-risk group for obstructive sleep apnea" according to the Berlin Questionnaire)
* Cardiovascular disease such as chronic heart failure
* Severe or untreated neurological diseases (e.g. Parkinson's disease, dementia, restless legs syndrome, narcolepsy)
* Alcohol and drug dependence
* Initiation of psychopharmacotherapy at a dosage provided for guideline-appropriate treatment of a mental disorder according to the Drug Compendium in the past 3 months
* Start of other psychotherapy procedures in the last 3 months
* Other parallel therapy methods (e.g. acupuncture, qigong, osteopathy)
* Somatic (sleep-disrupting) treatments, cortisone treatment, or radio-/chemotherapy in the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale (FSS) | The entire duration of the study is 3 years.
  The FSS comprises 9 questions, by answering which the patient can assess his limitations due to fatigue of the past week on a 7-point scale. The FSS is considered a well-established assessment tool for surveying subjective fatigue, the resulting limitations in daily, social, as well as occupational life and physical activities. Total score 36-52 is indicative of moderate fatigue ("mild/ no fatigue" at FSS total ≤ 35, "moderate fatigue" at 36 ≤ FSS total ≤ 52), score greater than or equal to 53 is indicative of severe fatigue ("severe fatigue" at FSS total ≥ 53).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland